CLINICAL TRIAL: NCT03169777
Title: NANT Colorectal Cancer (CRC) Vaccine: Combination Immunotherapy in Subjects With Recurrent or Metastatic CRC
Brief Title: QUILT-3.050: NANT Colorectal Cancer (CRC) Vaccine: Combination Immunotherapy in Subjects With Recurrent or Metastatic CRC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial not initiated
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.050
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — avelumab; Bevacizumab; Capecitabine; Cetuximab; Cyclophosphamide; Fluorouracil; Fulvestrant; Leucovorin; Taxes; Nivolumab; Omacor; Oxaliplatin; Radiosurgery; ALT-803; yeast-CEA vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nant CRC Vaccine (Experimental): avelumab, bevacizumab, capecitabine, cetuximab, cyclophosphamide, 5-fluorouracil, fulvestrant, leucovorin, nab paclitaxel, nivolumab, lovaza, oxaliplatin, stereotactic body radiation therapy, ALT-803, ETBX-011, ETBX-021, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, and haNK.
  Interventions: Biological: avelumab; Biological: bevacizumab; Drug: capecitabine; Biological: cetuximab; Drug: Cyclophosphamide; Drug: 5-Fluorouracil (5-FU); Drug: fulvestrant; Drug: leucovorin; Drug: nab paclitaxel; Biological: nivolumab; Drug: Lovaza; Drug: oxaliplatin; Radiation: Stereotactic Body Radiation Therapy; Biological: ALT-803; Biological: ETBX-011; Biological: ETBX-021; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-4000; Biological: GI-6207; Biological: GI-6301; Biological: haNK

INTERVENTIONS:
Biological: avelumab — Fully human anti-programmed death-ligand 1 (PD-L1) immunoglobulin (Ig)G1 lambda monoclonal antibody
Biological: bevacizumab — Recombinant human anti-vascular endothelial growth factor (VEGF) IgG1 monoclonal antibody
Drug: capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
Biological: cetuximab — Recombinant human/mouse chimeric anti-epidermal growth factor receptor (EGFR) IgG1 monoclonal antibody
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: 5-Fluorouracil (5-FU) — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
Drug: fulvestrant — 7-alpha-[9-(4,4,5,5,5-pentafluoropentylsulphinyl) nonyl]estra-1,3,5-(10)- triene-3,17-beta-diol
Drug: leucovorin — Calcium N-[p-[[[(6RS)-2-amino-5-formyl-5,6,7,8-tetrahydro-4-hydroxy-6-pteridinyl]methyl]amino]benzoyl]-L-glutamate (1:1)
Drug: nab paclitaxel — 5β,20-Epoxy-1,2α,4,7β,10β,13α-hexahydroxytax-11-en-9-one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)-N-benzoyl-3-phenylisoserine
Biological: nivolumab — Human anti-programmed cell death protein 1 (PD-1) IgG4 kappa monoclonal antibody
Drug: Lovaza — Omega-3-acid ethyl esters
Drug: oxaliplatin — cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum
Radiation: Stereotactic Body Radiation Therapy — (SBRT)
Biological: ALT-803 — recombinant human super agonist interleukin-15 (IL-15) complex
Biological: ETBX-011 — adenovirus serotype-5 [Ad5] [E1-, E2b-]-carcinoembryonic antigen [CEA] vaccine
Biological: ETBX-021 — Ad5 [E1-, E2b-]-human epidermal growth factor receptor 2 [HER2] vaccine
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury vaccine
Biological: ETBX-061 — Ad5 [E1-, E2b-]-mucin 1 [MUC1] vaccine
Biological: GI-4000 — RAS yeast vaccine
Biological: GI-6207 — CEA yeast vaccine
Biological: GI-6301 — Brachyury yeast vaccine
Biological: haNK — NK-92 [CD16.158V, ER IL-2], Suspension for Intravenous [IV] Infusion

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with recurrent and metastatic CRC.

DETAILED DESCRIPTION:
Treatment will be administered in 2 phases, an induction and a maintenance phase, as described below. Subjects will continue induction treatment for up to 1 year or until they experience progressive disease (PD) or unacceptable toxicity (not correctable with dose reduction), withdraw consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. Those who have a complete response (CR) in the induction phase will enter the maintenance phase of the study. Subjects may remain in the maintenance phase of the study for up to 1 year. Treatment will continue in the maintenance phase until the subject experiences PD or unacceptable toxicity (not correctable with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically confirmed recurrent or metastatic CRC.
4. ECOG performance status of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.5 cm.
6. Must have a recent tumor biopsy specimen obtained following the conclusion of the most recent anticancer treatment. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period.
7. Must be willing to provide blood samples and, if considered safe by the Investigator, a tumor biopsy specimen at 8 weeks after the start of treatment.
8. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
9. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment.

Exclusion Criteria:

1. History of persistent grade 2 or higher (CTCAE Version 4.03) hematologic toxicity resulting from previous therapy.
2. Within 5 years prior to first dose of study treatment, any evidence of other active malignancies or brain metastasis except for controlled basal cell carcinoma; prior history of in situ cancer (eg, breast, melanoma, and cervical); prior history of prostate cancer that is not under active systemic treatment (except hormonal therapy) and with undetectable PSA (< 0.2 ng/mL); and bulky (≥ 1.5 cm) disease with metastasis in the central hilar area of the chest and involving the pulmonary vasculature.
3. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
4. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, and autoimmune disease associated with lymphoma)
5. History of organ transplant requiring immunosuppression.
6. History of or active inflammatory bowel disease (eg, Crohn's disease and ulcerative colitis).
7. Requires whole blood transfusion to meet eligibility criteria.
8. Inadequate organ function, evidenced by the following laboratory results:

   1. WBC count < 2,500 cells/mm3
   2. Absolute neutrophil count < 1,500 cells/mm3.
   3. Platelet count < 100,000 cells/mm3.
   4. Hemoglobin < 9 g/dL.
   5. Total bilirubin greater than the ULN (unless the subject has documented Gilbert's syndrome).
   6. AST (SGOT) or ALT (SGPT) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   7. ALP levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   8. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   9. INR, aPTT, or PTT >1.5 × ULN (unless on therapeutic anti-coagulation).
9. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
10. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
11. Positive results of screening test for HIV, HBV, or HCV.
12. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
13. Known hypersensitivity to any component of the study medication(s).
14. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
15. Concurrent or prior use of a strong CYP3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
16. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
17. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
18. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
19. Concurrent participation in any interventional clinical trial.
20. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) and serious AEs (SAEs), graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. | 1 year
  Phase 1b primary endpoint (safety)
Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | 1 year
  Phase 2 primary endpoint (ORR by RECIST)
ORR by Immune-related response criteria (irRC ) | 1 year
  Phase 2 primary endpoint (ORR by irRC)

SECONDARY OUTCOMES:
ORR by RECIST Version 1.1 | 1 year
  Phase 1b secondary endpoint (ORR by RECIST)
ORR by irRC | 1 year
  Phase 1b secondary endpoint (ORR by irRC)
Progression-free survival (PFS) by RECIST Version 1.1 | 2 year
  Phase 1b and 2 secondary endpoint (PFS by RECIST)
PFS by irRC | 2 years
  Phase 1b and 2 secondary endpoint (PFS by irRC)
Overall survival (OS): time from the date of first treatment to the date of death (any cause) | 2 years
  Phase 1b and 2 secondary endpoint (OS)
Duration of response (DR): time from the date of first response (partial response (PR) or complete response (CR)) to the date of disease progression or death (any cause) whichever occurs first | 2 years
  Phase 1b and 2 secondary endpoint (DR)
Disease control rate (DCR): confirmed complete response, partial response, or stable disease lasting for at least 2 months | 2 months
  Phase 1b and 2 secondary endpoint (DCR)
Quality of life (QoL) by patient-reported outcome using the Functional Assessment of Cancer Therapy-Colorectal Cancer (FACT-C) questionnaire | 2 years
  Phase 1b and 2 secondary endpoint (QoL)
Incidence of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs), graded using the NCI CTCAE Version 4.03 | 1 year
  Phase 2 secondary endpoint (AEs)

IPD SHARING:
Plan to Share IPD: No